CLINICAL TRIAL: NCT06245772
Title: A National, Multicentre, Non-interventional, Prospective, Longitudinal Study to Assess CARegiver BURden, Effectiveness and Other Health Care Measures on Functional Disability, in Patients Treated With Abobotulinumtoxin A for Upper Limb Spasticity in Routine Clinical Practice.
Brief Title: CARegiver BURden, Effectiveness and Other Health Care Measures on Functional Disability, in Patients Treated With Abobotulinumtoxin A for Upper Limb Spasticity
Acronym: CARBUR
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52120-459
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Upper Limb Injury
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to perform, in real world clinical practice, a three-dimensional assessment from patient's, caregiver's and physician's perspectives, of the impact of AboBoNT-A on caregiver burden, functional disability and other health care measures in patients affected with ULS due to acquired brain injuries.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able to comply with the protocol;
2. Male and female patients who are at least 18 years old;
3. The patient is supported by an identified caregiver (family member or other nonpaid adult

   - if the patient has more than one caregiver, the main caregiver will be selected) who provides daily supervision or direct assistance to the care recipient;
4. The patient has been diagnosed with ULS due to non-progressive acquired brain injuries (stroke, traumatic brain injury, surgical resection of non-progressive tumours, other) or due to non-progressive spinal cord injury with stability of spasticity of the upper limbs;
5. The decision to treat the patient with AboBoNT-A by the care provider will be made prior to, and independently from the decision to enrol the patient in the observational study;
6. The patient is covered by a healthcare insurance;
7. The cognitive and health status of the patient is compatible with the participation to the study.

For Caregivers :

(8) The caregiver is able to comply with the protocol; (9) Male and female caregivers who are at least 18 years old; (10) The cognitive and health status of the caregiver is compatible with the participation to the study.

Exclusion Criteria:

1. Contraindication to BoNT-A treatment;
2. Previously treated with BoNT-A in upper limbs within the last 12 months;
3. Patients and if applicable Legally Authorized Representative (LAR) of patient under curatorship or deprived of liberty who are opposed to their data collection
4. Caregivers who are opposed to their data collection;
5. Caregivers already included for another patient;
6. Current participation in any other interventional clinical study or have participated within the 12 weeks prior to the inclusion visit;
7. Non-ambulatory patients except for those who have been hospitalized for the purpose of their BoNT-A injection (maximum length of stay as per clinical judgment of the investigator);
8. Vulnerable patients (i.e. pregnant and/or lactating women, children, patient under curatorship or deprived of liberty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ULS who will start AboBoNT-A treatment in upper limbs as part of routine clinical practice should be recruited. Patients who received BoNT-A injections in upper limbs less than one year prior to inclusion should not be included in the study. Patients who previously received BoNTA injections in body parts other than upper limbs could be included in the study, regardless of injection anteriority.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the 5-item Carer Burden Scale (CBS) mean score | From baseline to 8 weeks
  The 5-item Carer Burden Scale is 5-point Likert scale ranging from 0 (no difficulty) to 4 (cannot complete the task), so that higher scores indicate greater burden.

SECONDARY OUTCOMES:
Patient's demographic data | through study completion, an average of 14 months
  Patient's Characteristics
Caregiver's demographic data; | through study completion, an average of 14 months
  Patient's Characteristics
Aetiology of spasticity; | through study completion, an average of 14 months
  Patient's Characteristics
Affected upper limb | through study completion, an average of 14 months
  Patient's Characteristics
Ascribed spastic muscle group(s); | through study completion, an average of 14 months
  Patient's Characteristics
Time since onset of the aetiology of upper limb spasticity (ULS) | through study completion, an average of 14 months
  Patient's Characteristics
Associated lower limb spasticity (LLS) | through study completion, an average of 14 months
  Patient's Characteristics
Global autonomy evaluation (modified Rankin Scale). | through study completion, an average of 14 months
  Patient's Characteristics
Total dose injected in ULS per cycle; | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Dose per muscle group; | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Number of injected muscle group(s) | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Injections Practices - Total dose injected per cycle (any indication); | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Time between two injections; | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Criteria for reinjection; | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Reasons for treatment discontinuation, if any, and subsequent therapy if any. | through study completion, an average of 14 months
  Injections Practices; over a period of 3 cycles of treatment with AboBoNT-A in patients affected with ULS.
Change from baseline in Carer Burden Scale (CBS) | through study completion, an average of 14 months
  Caregiver Burden; The impact of treatment on the physical burden of the caregiver will be assessed by the same caregiver using a modified paper version of the CBS self-administered questionnaire
Change from baseline in ZBI-12 total score to the end of each AboBoNT-A cycle | through study completion, an average of 14 months
  Treatment Effectiveness; ZBI-12 is a self-administered questionnaire for measuring caregiving burden
Goal score | through study completion, an average of 14 months
  Treatment Effectiveness; To assess goals achievement it will be used an adapted scale / Therapeutic Goal Attainment Scaling (TGAS) with pre-defined goals
Goal score change | through study completion, an average of 14 months
  Treatment Effectiveness; To assess goals achievement it will be used an adapted scale / Therapeutic Goal Attainment Scaling (TGAS) with pre-defined goals
Distribution of Goals each AboBoNT-A cycle; | through study completion, an average of 26 months
  Treatment Effectiveness; To assess goals achievement it will be used an adapted scale / Therapeutic Goal Attainment Scaling (TGAS) with pre-defined goals
Proportion of patients "attaining" the primary Goal | through study completion, an average of 14 months
  Treatment Effectiveness
Proportion of patients "attaining" at least one Goal | through study completion, an average of 14 months
  Treatment Effectiveness; To assess goals achievement it will be used an adapted scale / Therapeutic Goal Attainment Scaling (TGAS) with pre-defined goals
Proportion of patients "attaining" the pre-defined goal | through study completion, an average of 14 months
  Treatment Effectiveness; To assess goals achievement it will be used an adapted scale / Therapeutic Goal Attainment Scaling (TGAS) with pre-defined goals
Change from baseline in Modified Ashworth Scale (MAS) score. | through study completion, an average of 14 months
  Treatment Effectiveness; Based on routine clinical examination, group muscle tone assessments performed by the Investigator according to the MAS will be recorded
Change from baseline in SQoL-6D total score | through study completion, an average of 14 months
  Patient's Spasticity-Related Health Status (PS-RHS); The SQoL-6D consists of a 6-dimensions self-administered questionnaire that provides an overall picture of ULS spasticity-related health status
Change from baseline in SQoL-6D pain/discomfort subscore | through study completion, an average of 14 months
  Patient's Spasticity-Related Health Status (PS-RHS); The SQoL-6D consists of a 6-dimensions self-administered questionnaire that provides an overall picture of ULS spasticity-related health status
Number and percentage of patients with the following concomitant medications: oral antispasticity medications, pain medications (nociceptive and neuropathic pain), psychotropic drugs and anticoagulant drugs. | Up to 14 months
  Concomitant Medications, Non-Drug Therapies and Surgeries
Number and percentage of patients with the following concomitant non-drug therapies for the management of ULS: physiotherapy and use of orthoses; | Up to 14 months
  Concomitant Medications, Non-Drug Therapies and Surgeries
Number and percentage of patients with concomitant surgical procedures impacting caregivers' burden and patients' health. | Up to 14 months
  Concomitant Medications, Non-Drug Therapies and Surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (37):
- France (37):
  - CH Bagnères, Bagnères-de-Bigorre
  - CH Bar le Duc, Bar-le-Duc
  - Besançon - CHU/CRRF de Bréguille/Salin les bains, Besançon
  - CHU Bordeaux - Hopital Tastet-Girard, Bordeaux
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CHU Brest, Brest
  - SSR Tour de Gassies, Bruges
  - CH Colmar, Colmar
  - Centre de rééducation des 3 vallées, Corbie
  - CH Dax, Dax
  - CRF DIivio Dijon, Dijon
  - Fondation hopale - Fouqière-lez-Lens, Fouquières-lès-Lens
  - Clinique de Verdaich, Gaillac-Toulza
  - Garches, Garche
  - Groupe Hospitalier De Gonesse, Gonesse
  - HCL - Renée Sabran, Hyères
  - Crf Bel Air, La Membrolle-sur-Choisille
  - CHU Lille, Lille
  - Clinique Saint Martin Sud, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - Hôpital Rothschild, Paris
  - Ste Anne, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Pole St Hélier, Rennes
  - Fondation Ildys - Roscoff, Roscoff
  - CH Saint Denis, Saint-Denis
  - SSR Val Rosay UGECAM, Saint-Didier-au-Mont-d'Or
  - CH Ariège Couserans Site de Rozès, Saint-Girons
  - CH Saint Jean de Luz, Saint-Jean-de-Luz
  - Le Centre Médical Germaine Revel, Saint-Maurice-sur-Dargoire
  - CHU Amiens, Salouël
  - CHU Toulouse, Toulouse
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/